CLINICAL TRIAL: NCT02156986
Title: Effect of Food Structural Properties on Infants and Toddlers Mastication Abilities
Brief Title: Chewing Capability Study for Infants and Toddlers
Status: Completed | Type: Observational
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Other Study IDs: 13.03.INF
Record Dates: First submitted 2014-06-04; First posted 2014-06-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Healthy

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 9 month old infant
- 12 month old infant
- 18 month old toddler
- 24 month old toddler
- 36 month old toddler

SUMMARY:
The main objective of the study is to conduct a pilot study on the characterization of the mastication abilities of infants and toddlers using different commercial cereal based products in order to gain knowledge and be able to plan future studies.

ELIGIBILITY:
Inclusion Criteria:

* Born at term (37+ weeks)
* Familiar with solid foods
* No known history of food allergies
* Child must be within 2 weeks of the targeted age group for 9 months, within 1 month for 12 months, within 2 months for 18 and 24 months, and within 3 months for 36 months for this study.
* English must be the primary language of the participant and family.
* Having obtained his/her caregiver's or legal representative's informed consent.

Exclusion Criteria:

* History of speech/language, cognitive, or physical impairments as indicated on the self-reported medical history questionnaire completed by caregiver or legal guardian
* Any previously undiagnosed speech/language or cognitive impairment detected by the Investigator. In the case a subject is identified as being at risk for a communication or feeding impairment, the caregiver will be notified and provided with a list of local speech-language pathology providers who could perform a formal assessment
* History of poor weight gain/ weight loss, food allergies, difficulties with sucking, difficulties with chewing and/ or swallowing, frequent drooling (for age groups 18, 24, and 36 months), frequent choking, gastro-esophageal reflux, frequent spitting up/ vomiting (for age groups 18, 24, and 36 months) or irritability after feedings/ eating
* Latex allergies
* Currently participating in or having participated in a similar clinical trial related to food/diet within the last 9 months
* Caregiver must not be under the age of 18 years old.

Ages: 9 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The subjects investigated will be healthy infants and toddlers ranging from 9 to 36 months in 5 groups:
  * 9 months (±2 weeks),
  * 12 months (±1 month),
  * 18 months (±2 months),
  * 24 months (±2 months),
  * 36 months (±3 months).
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Muscle activities involved in the mastication using Electromyography (EMG) | One day during the study visit 2

CONTACTS AND LOCATIONS:
Locations (1):
- MGH Institute of Health Professions, Boston, Massachusetts, United States